CLINICAL TRIAL: NCT00174005
Title: Validity and Reliability in Measuring Tendon and Muscular Morphologic Characteristics of Biceps and Triceps by Using Ultrasound
Brief Title: Validity and Reliability in Measuring Biceps and Triceps by Using Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701181
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 1994-12

CONDITIONS: Healthy
Keywords: muscle; tendon

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to estimate the validity and reliability in the measurement of bicep and tricep tendons and muscular morphologic characteristics by using ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age range from 19-35 years

Exclusion Criteria:

* History of shoulder or elbow pain which needs medical treatment or surgery

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Kuo Wang, PhD, Study Director — School and Graduate Institute of Physical Therapy, National Taiwan University; Hsing-Kuo Wang, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan